CLINICAL TRIAL: NCT01692509
Title: Observation of Non Invasive Ventilation (NIV) Related Practices, Monitoring of the NIV Treatment Effect and of the Patient's Comfort During NIV
Brief Title: Non Invasive Ventilation (NIV) Related Practices, Monitoring of the NIV Treatment Effect and of the Patient's Comfort
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Prof. Philippe Jolliet, Main investigator, University of Lausanne Hospitals
Other Study IDs: NIV related practices
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Respiratory Failure Requiring Non Invasive Ventilation
Keywords: Non invasive ventilation; Respiratory failure; Respiratory comfort
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients requiring NIV: Patients requiring NIV because of acute respiratory failure

SUMMARY:
The practices and processes related to the administration of noninvasive ventilation (NIV) in the adult intensive care unit (ICU) of the University hospital of Lausanne will be recorded by an investigator at the bedside. The effect of the NIV treatment on various respiratory parameters ( respiratory rate, expired tidal volume, minute ventilation) will also be recorded using a pneumotachograph. Finally patient's comfort during NIV treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory failure
* Therapeutic treatment by NIV required

Exclusion Criteria:

* Age < 18 years old
* Prophylactic NIV treatment
* Continuous Positive Airway Pressure (CPAP)treatment
* Denied consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized in the CHUV intensive care unit who require non invasive ventilation because of respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Documentation of practices and processes related to NIV treatment
  Documentation of practices and processes related to NIV administration in the adult intensive care unit(type of ventilator used, type of interface chosen, initial settings, organization of the care team and interactions between caregivers).

SECONDARY OUTCOMES:
Patient's Respiratory comfort
  Patient's respiratory comfort during NIV will be assessed both by the patients themselves with a visual analogic scale and by the investigator.
Ventilatory parameters
  Tidal volume, respiratory rate, inspiratory time, expiratory time and maximal and mean airway pressure will be measured from the continuous recording of airway pressure and flow obtained with a pneumotachograph.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jolliet, Professor, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Intensive care and burn unit, University Hospital of Lausanne, Lausanne, Switzerland